CLINICAL TRIAL: NCT02275312
Title: ETREAT: A Prospective Observational Study to Evaluate the Effectiveness of Botulinum Toxin Type A (BoNT-A) Injections in Patients With Post-stroke Upper and/or Lower Limb Spasticity in the Early Stage of Spasticity Development.
Brief Title: ETREAT Study on Effectiveness of Botulinum Toxin Type A Injections to Treat Post-stroke Upper and/or Lower Limb Spasticity
Acronym: ETREAT
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-92-52120-192
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Spasticity
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to evaluate the effectiveness of BoNT-A on functional improvement in patients with post-stroke upper and/or lower limb spasticity in the early stage of spasticity development, according to routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18-80 years.
* Poststroke limb spasticity.
* Patients who have suffered a stroke in the previous 6 months.
* Treatment goal has been previously agreed with the patient or their legal representative.
* Patients with clinically significant poststroke upper/lower limb spasticity, in whom it has been decided to perform multidisciplinary treatment with BoNT-A + rehabilitation.
* No previous treatment with BoNT-A.
* Patient is able to follow the protocol.
* Written informed consent.

Exclusion Criteria:

* Neuromuscular disease.
* Use of drugs that interfere with neuromuscular transmission.
* Any other condition that could interfere with rehabilitation or evaluation of the results.
* Diagnosis of spasticity not associated with stroke.
* Pregnant or nursing mothers.
* Prior participation in any other study in the 6 months before study entry

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-stroke spasticity
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in Goal Attainment Scale (GAS) score. | Baseline, 16 months

SECONDARY OUTCOMES:
Spasticity patterns will be defined in patients with upper and/or lower limb spasticity in the early stage after stroke | Baseline, 16 months
  Descriptive statistics will be presented in addition to 95% confidence intervals for the mean and percentages
Change in Modified Ashworth Scale (MAS) score. | Baseline, 16 months
Baseline characteristics of patients | Baseline
  Demographic characteristics
Percentage of patients reporting functional improvement evaluated by Goal Attainment Scale (GAS) score. | From baseline up to 16 months
Change in pain according to Visual Analog Scale (VAS). | Baseline, 16 months
Passive function of upper and/or lower limbs according to primary treatment target (PTT) from the disability assessment scale (DAS). | Baseline, 16 months
Comfortable barefoot walking speed, measured with the 10-meter walking speed test. | Baseline, 16 months
Change on EQ-5D quality of life questionnaire | Baseline, 16 months
Estimation of use of healthcare resources and costs associated with management of spasticity. | From baseline up to 16 months
Time interval between injections | From baseline up to 16 months
Cost per patient | From baseline up to 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (17):
- Spain (17):
  - Barcelona
  - Bilbao
  - Cadiz
  - Córdoba
  - Granada
  - Huelva
  - Las Palmas de Gran Canaria
  - Lleida
  - Madrid
  - Murcia
  - Palma de Mallorca
  - Pontevedra
  - Salamanca
  - San Sebastián
  - Santiago
  - Seville
  - Valladolid